CLINICAL TRIAL: NCT00507104
Title: Prospective Longitudinal Study on Pituitary Functions After TBI and/or SAH
Brief Title: Pituitary Functions After Traumatic Brain Injury (TBI) and/or Subarachnoid Hemorrhage (SAH)
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: pitfunction_TBI_SAH
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage; Hypopituitarism
Keywords: traumatic brain injury; Subarachnoid Hemorrhage; Hypopituitarism
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Hypopituitarism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study performs assessments of pituitary functions by basal hormone levels in the acute phase after TBI and/or SAH followed by detailed endocrine tests (insulin-induced hypoglycemia or growth hormone releasing hormone-arginine-corticotropin releasing hormone-leuteinizing hormone releasing hormone [GHRH-arginine-CRH-LHRH] test) after 4 and 12 months.

DETAILED DESCRIPTION:
Recent data have demonstrated that hypopituitarism seems to be a frequent finding after traumatic brain injury (TBI) and/or subarachnoid hemorrhage (SAH). However, most of these studies referred to retrospective evaluations. There are only few prospective data, and no longitudinal study routinely taking into account the assessment of anterior pituitary function in the acute phase after TBI or SAH so far.

We prospectively evaluate pituitary functions in patients in the acute phase after TBI or SAH and a control group of patients with trauma not involving the brain. Endocrine data included basal anterior pituitary lobe hormone, IGF-1 and testosterone serum levels (Immulite 2000) within the first 8 hours after TBI or SAH. Further endocrine evaluation was performed by means of either a combined GHRH-arginine-CRH-LHRH test or an insulin-induced hypoglycemia test after 4 months and 12 months. To rule out an assay related bias with regard to GH and IGF-1, all hormone levels were cross-checked by a supersensitive assay in another laboratory.

ELIGIBILITY:
Inclusion Criteria:

* TBI or SAH
* Control group: injury without involvement of the brain/skull

Exclusion Criteria:

* Pregnancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Buchfelder, M.D., Ph.D., Study Chair — Department of Neurosurgery, University of Erlangen; Juergen Kreutzer, M.D., Principal Investigator — Department of Neurosurgery, University of Erlangen; Christioph Schöfl, M.D., Ph.D., Principal Investigator — Department of Neurosurgery, Division Neuroendocrinology, University of Erlangen; Andrea Kleindienst, M.D., Principal Investigator — Department of Neurosurgery, University of Erlangen
Locations (1):
- Department of Neurosurgery, University of Erlangen, Erlangen, Germany